CLINICAL TRIAL: NCT05196451
Title: Short-time Behavioural Intervention in Post-Covid Syndrome (SIPCOV): A Pragmatic Randomised Controlled Trial
Brief Title: Short-time Intervention in Post-Covid Syndrome Syndrome (SIPCOV): A Pragmatic Randomised Controlled Trial
Acronym: SIPCOV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Akershus (Other)
Responsible Party: Principal Investigator, Vegard Wyller, Professor, University Hospital, Akershus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 21/12248
Record Dates: First submitted 2022-01-14; First posted 2022-01-19 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short-time rehabilitation (Active Comparator): The intervention consists of an individualized numbers of outpatient encounters (min. 2, max. 8) with medical doctors and physiotherapists at Kysthospitalet, Stavern, Norway. The encounters aim to foster a rehabilitation process based upon principles from Cognitive Behavioral Therapy (CBT)
  Interventions: Behavioral: Rehabilitation based on CBT principles
- Care as usual (No Intervention)

INTERVENTIONS:
Behavioral: Rehabilitation based on CBT principles — Cf. arm description
  Arms: Short-time rehabilitation

SUMMARY:
The present study is a 2-arm pragmatic randomised controlled trial (RCT) in which 310 patients who suffer from post-Covid syndrome are randomised to either a short-time outpatient-based rehabilitation program (the intervention) or care as usual in a 1:1 ratio. Assessments will take place immediately before randomisation (T0), after intervention or care as usual (T1), and 6 months after T1 (T2). Patients will be recruited from General Practitioners (GP's) as well as social media and self-referral to the involved institutions.

ELIGIBILITY:
Inclusion Criteria:

* Fulfils pragmatic diagnostic criteria of idiopathic post-Covid syndrome: a) Confirmed acute Covid-19 by a positive PCR for SARS-CoV-2; b) Persistent symptoms at least 3 months following acute Covid-19 without symptom-free interval; c) Functional disability to an extent that interrupts all or a majority of normal activities (such as work/school attendance, physical exercise, social activities, etc.)
* Lives in one of the following Norwegian counties: Oslo, Viken, Innlandet, Vestfold og Telemark, Agder
* Informed consent to participation

Exclusion criteria

* Other chronic illnesses or demanding life situations that might explain persistent symptoms and disability
* Sustained organ damage (lung, heart, brain) following acute, serious Covid-19
* Bedridden
* Insufficient command of Norwegian language

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 314 (Actual)
Dates: Start 2022-02-21 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Physical Functioning | Immediately after intervention (time T1)
  Physical Functioning subscale from the SF-36 inventory. The SF-36 comprises a total of 36 items on subjective mental, social and physical health, which are assigned to 8 dimensions. Scale ranging from 0 (poor quality of life) to 100 (best)

SECONDARY OUTCOMES:
Fatigue | Immediately after intervention (time T1)
  Chalder Fatigue Questionnaire (CFQ), total sum score. Range from 0-33, higher scores means more fatigue.
Fatigue | At 12 months follow-up (time T2)
  Chalder fatigue questionnaire, total sum score
Depression/anxiety | Immediately after intervention (time T1)
  Hospital Anxiety and Depresssion Scale, total score. Higher scores means more depression/anxiety symptoms.
Depression/anxiety | At 12 months follow-up (time T2)
  Hospital Anxiety and Depresssion Scale, total score
Adverse effects | Immediately after intervention (time T1)
  Self-invented questionnaire on adverse effects
Adverse effects | At 12 months follow-up (time T2)
  Self-invented questionnaire on adverse effects
Physical Functioning | At 12 months follow-up (time T2)
  Physical Functioning subscale from the SF-36 inventory
Recovery from PIFS | Immediately after intervention (time T1)
  Recovery from post-infective fatigue syndrome (PIFS)
Recovery from PIFS | At 12 months follow-up (time T2)
  Recovery from post-infective fatigue syndrome (PIFS)

CONTACTS AND LOCATIONS:
Overall Officials: Vegard B Wyller, Principal Investigator — University Hospital, Akershus
Locations (1):
- Vegard Bratholm Wyller, Oslo, Norway

REFERENCES:
- [Derived] Nerli TF, Selvakumar J, Cvejic E, Heier I, Pedersen M, Johnsen TL, Wyller VBB. Brief Outpatient Rehabilitation Program for Post-COVID-19 Condition: A Randomized Clinical Trial. JAMA Netw Open. 2024 Dec 2;7(12):e2450744. doi: 10.1001/jamanetworkopen.2024.50744. PMID 39699896

DOCUMENTS (2):
  • Study Protocol (2022-02-20): https://cdn.clinicaltrials.gov/large-docs/51/NCT05196451/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-23): https://cdn.clinicaltrials.gov/large-docs/51/NCT05196451/SAP_001.pdf